CLINICAL TRIAL: NCT00447148
Title: Standard vs. 3-Dimensional Coronary Angiography: a Paired Comparison Using Intra-Coronary Marker Wires as Matched-Comparison "Gold Standard"
Brief Title: Standard vs. 3-Dimensional Coronary Angiography: a Paired Comparison
Acronym: 3-DCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antwerp Cardiovascular Institute Middelheim (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACIM 2006-001
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): Paired comparison of 2 angiographic techniques
  Interventions: Procedure: 3-dimensional coronary angiography

INTERVENTIONS:
Procedure: 3-dimensional coronary angiography — 3-dimensional coronary angiography
  Other Names: coronary angiography

SUMMARY:
Aim of this study is to evaluate whether the length of coronary segments, assessed by an experienced operator, using the "optimal view" of standard 2-dimensional coronary angiography, is over/underestimated with respect to the one evaluated automatically with the help of a 3-dimensional coronary reconstruction model. Moreover, both techniques are compared with an "in-vivo" surrogate of the real length of the coronary segment under evaluation, i.e. an intra-coronary marker guide-wire, which is a wire with markers placed at fixed and known distance along its length in its distal (intra-coronary) part. Two hypotheses are tested: (1) the length of a coronary segment evaluated with a standard 2-dimensional "optimal view" over/underestimates the length assessed by a 3-dimensional coronary model that automatically detects the least foreshortened length of the segment under evaluation, and (2) the 3-dimensional model approximates more closely than standard 2-dimensional angiography, the real length of the segment detected by the marker guide-wire.

DETAILED DESCRIPTION:
The potential to improve the accuracy of the assessment of the coronary tree by means of 3-D modeling reconstruction may lead to an evaluation of the coronary artery anatomy that approximates more correctly the real anatomy, thus subsequently leading to a more tailored diagnosis and therapy for the patients with ischemic heart disease.

Aim of the current study is to assess whether a 3-D model of the coronary tree offers a less foreshortened and less operator-dependent evaluation of the length of the coronary arteries with respect to standard coronary angiography. Furthermore, for the first time "in-vivo", a comparison with the "real" length of the vessel will be performed using as "gold standard" an intra-coronary guide-wire with radiopaque markers at fixed and known distance one from the other along its distal part.

ELIGIBILITY:
Inclusion Criteria:

Clinical

* Age > 18 years.
* Ability to give informed consent.
* Clinical evidence of coronary artery disease:

  * recent (< 72 hours) acute myocardial infarction,
  * stable angina with documented positive stress test,
  * unstable angina with documented ischemia (positive ECG or troponin test or documented positive stress test).

Angiographic

* Eligibility for PCI in at least one de-novo stenosis in a native coronary artery, after the index angiogram.
* Planned PCI according to a previous coronary angiogram.

Exclusion Criteria:

Clinical

* Pregnancy.
* Chronic or acute renal failure (serum creatinine > 1.8 mg/dL or hemodialysis).
* Urgent procedure (a procedure carried out before the next referring day, for example for acute myocardial infarction, unstable angina refractory to medical therapy or cardiogenic shock).
* Contraindications or known hypersensitivity to contrast media.
* Enrollment in another study protocol.

Angiographic

* Significant left main coronary artery disease.
* PCI for a total occlusion of a major coronary vessel (LAD, LCX or RCA).
* Extensive thrombotic burden in a coronary lesion (thrombus grade 3/4).
* TIMI flow <3 distal to the lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
standard coronary angiography over/underestimates the length of the coronary segment evaluated. | peri-procedural

SECONDARY OUTCOMES:
The length of the segments, evaluated with standard and 3-D angiography, will be compared with the length of the segment measured with the marker guide-wire.
Each group of the same vessel(LAD, RCA, CX) will be evaluated separately.
All the QCA results of standard angiography will be compared with those of 3-D angiography, in particular in the segments where the lesion is.
The percentage of vessel foreshortening of the standard angiography operator-selected "working view" will be compared to the least foreshortened view automatically selected with the 3-D angiography reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Agostoni, MD, Principal Investigator — Antwerp Cardiovascular Institute Middelheim; Stefan Verheye, MD, PhD, Study Chair — Antwerp Cardiovascular Institute Middelheim; Glenn Van Langenhove, MD, PhD, Study Director — Antwerp Cardiovascular Institute Middelheim
Locations (1):
- Antwerp Cardiovascular Institute Middelheim, Antwerp, Belgium